CLINICAL TRIAL: NCT00897533
Title: Development of a Model to Predict Progression Free Survival After Treatment With Erlotinib in E3503
Brief Title: Development of a Model to Predict Progression-Free Survival After Erlotinib in Patients With Non-Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000543981; ECOG-E3503T1
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung; squamous cell lung cancer; bronchoalveolar cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Chromosome Mapping; Amplified Fragment Length Polymorphism Analysis; Immunohistochemistry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: gene mapping
Genetic: polymorphism analysis
Other: diagnostic laboratory biomarker analysis
Other: immunohistochemistry staining method

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients respond to treatment with erlotinib.

PURPOSE: This laboratory study is developing a model to predict progression-free survival after erlotinib in patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess mesenchymal and epithelial markers in tissues from patients with non-small cell lung cancer treated with erlotinib hydrochloride on clinical trial ECOG-E3503.
* Determine the loss of epithelial markers (E-cadherin) and gain of mesenchymal markers (vimentin/cytokeratin co-expression) in these patients.
* Assess whether mesenchymal and epithelial markers are predictive of progression-free survival (PFS) of these patients.
* Identify a single nucleotide polymorphism profile via whole genome mapping and other known biomarkers to predict PFS of these patients.

OUTLINE: Tissue samples are analyzed by whole genome mapping for single nucleotide polymorphism (SNP) rate and by signal detection rate and by quantitative immunohistochemistry for mesenchymal (vimentin/cytokeratin) and epithelial (E-cadherin) marker transitions. After biomarker identification and gene mapping are complete, a model to predict progression-free survival in these patients is developed.

PROJECTED ACCRUAL: A total of 137 samples will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of non-small cell lung cancer, including any of the following subtypes:

  * Adenocarcinoma
  * Squamous cell carcinoma
  * Bronchoalveolar carcinoma
  * Carcinoid
* Stage IIIB or IV or recurrent disease
* Must have received treatment with erlotinib hydrochloride on clinical trial ECOG-E3503

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Samples submitted for research from patients participating in E3503
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2007-04-13 (Actual); Primary Completion 2008-04-13 (Actual); Study Completion 2008-04-13 (Actual)

PRIMARY OUTCOMES:
Mesenchymal and epithelial markers | 1 month
  Mesenchymal and epithelial markers
Loss of epithelial markers (E-cadherin) and gain of mesenchymal markers (vimentin/cytokeratin co-expression) | 1 month
  Loss of epithelial markers (E-cadherin) and gain of mesenchymal markers
Correlation of progression-free survival (PFS) by mesenchymal and epithelial markers | 1 month
  Correlation of progression-free survival (PFS) by mesenchymal and epithelial markers
Identification of a single nucleotide polymorphism profile via whole genome mapping and other known biomarkers to predict PFS | 1 month
  Identification of a single nucleotide polymorphism profile via whole genome mapping and other known biomarkers to predict PFS

CONTACTS AND LOCATIONS:
Overall Officials: Jill Kolesar, PharmD, Study Chair — University of Wisconsin, Madison

REFERENCES:
- [Result] Amann JM, Lee JW, Roder H, Brahmer J, Gonzalez A, Schiller JH, Carbone DP. Genetic and proteomic features associated with survival after treatment with erlotinib in first-line therapy of non-small cell lung cancer in Eastern Cooperative Oncology Group 3503. J Thorac Oncol. 2010 Feb;5(2):169-78. doi: 10.1097/JTO.0b013e3181c8cbd9. PMID 20035238